CLINICAL TRIAL: NCT02980809
Title: Topotecan Plus Apatinib Versus Topotecan Alone as Second-line Therapy in Small-cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Hospitals affiliated to the China PLA General Hospital (Other Government)
Responsible Party: Principal Investigator, Min-hang Zhou, doctor, First Hospitals affiliated to the China PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: gsk-001
Record Dates: First submitted 2016-11-24; First posted 2016-12-02 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — apatinib; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apatinib and topotecan (Experimental): Patients receive IV topotecan 1.5 mg/m2/d on days 1 through 5, apatinib 250mg/d, every 21 days, until disease progression.
  Interventions: Drug: Apatinib; Drug: Topotecan
- Topotecan (Placebo Comparator): Patients receive IV topotecan 1.5 mg/m2/d on days 1 through 5 every 21 days, until disease progression.
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Apatinib
  Arms: Apatinib and topotecan
Drug: Topotecan

SUMMARY:
The purpose of this study is to determine whether topotecan plus apatinib are superior to topotecan alone as second-line therapy in small-cell lung cancer.

DETAILED DESCRIPTION:
Small-cell lung cancer (SCLC) is an aggressive tumor and most patients experienced relapse or progression after standard chemotherapy. Topotecan is active as second-line therapy for SCLC patients. However, even in sensitive patients, only 20% response rate and a median time to progression of 12 weeks are observed. New therapeutic options in SCLC are needed. Apatinib is a small-molecule tyrosine kinase inhibitor that inhibits vascular endothelial growth factor receptor 2. It has been approved in patients with advanced gastric cancer refractory to two or more lines of prior chemotherapy. The efficacy of apatinib in SCLC is unknown. The purpose of this study is to determine whether topotecan plus apatinib are superior to topotecan alone as second-line therapy in small-cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* limited or extensive-stage SCLC who had failed to first-line therapy
* ≥18 years old
* Eastern Cooperative Oncology Group performance status ≤2
* at least one measurable lesion as defined by RECIST (version 1.1)
* at least one measurable lung tumor lesion
* WBC count ≥3,500/μL, neutrophils ≥1,500μL, platelets ≥100,000μL, hemoglobin ≥ 9.0 g/dL
* AST, and ALT ≤2 × the upper limit of normal or ≤5 × the upper limit of normal with liver metastases.

Exclusion Criteria:

* symptomatic CNS metastases
* concomitant or previous malignancies within the last 5 years
* severe comorbidities; prior topotecan therapy
* hypersensitivity or other contraindication to the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-03; Primary Completion 2019-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 1 year

SECONDARY OUTCOMES:
Response rate | 1 year
Toxicity assessed by common terminology criteria for adverse events(CTCAE) V4.0 | 1 year
  Toxicity is assessed by common terminology criteria for adverse events(CTCAE) V4.0

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] O'Brien ME, Ciuleanu TE, Tsekov H, Shparyk Y, Cucevia B, Juhasz G, Thatcher N, Ross GA, Dane GC, Crofts T. Phase III trial comparing supportive care alone with supportive care with oral topotecan in patients with relapsed small-cell lung cancer. J Clin Oncol. 2006 Dec 1;24(34):5441-7. doi: 10.1200/JCO.2006.06.5821. PMID 17135646
- [Background] Eckardt JR, von Pawel J, Pujol JL, Papai Z, Quoix E, Ardizzoni A, Poulin R, Preston AJ, Dane G, Ross G. Phase III study of oral compared with intravenous topotecan as second-line therapy in small-cell lung cancer. J Clin Oncol. 2007 May 20;25(15):2086-92. doi: 10.1200/JCO.2006.08.3998. PMID 17513814
- [Background] Li J, Qin S, Xu J, Xiong J, Wu C, Bai Y, Liu W, Tong J, Liu Y, Xu R, Wang Z, Wang Q, Ouyang X, Yang Y, Ba Y, Liang J, Lin X, Luo D, Zheng R, Wang X, Sun G, Wang L, Zheng L, Guo H, Wu J, Xu N, Yang J, Zhang H, Cheng Y, Wang N, Chen L, Fan Z, Sun P, Yu H. Randomized, Double-Blind, Placebo-Controlled Phase III Trial of Apatinib in Patients With Chemotherapy-Refractory Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction. J Clin Oncol. 2016 May 1;34(13):1448-54. doi: 10.1200/JCO.2015.63.5995. Epub 2016 Feb 16. PMID 26884585
- [Background] Fruh M, De Ruysscher D, Popat S, Crino L, Peters S, Felip E; ESMO Guidelines Working Group. Small-cell lung cancer (SCLC): ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2013 Oct;24 Suppl 6:vi99-105. doi: 10.1093/annonc/mdt178. Epub 2013 Jun 27. No abstract available. PMID 23813929